CLINICAL TRIAL: NCT03488329
Title: Effect of Nutritional Efforts on Discharged Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Jonas Anias Svendsen, Research Associate, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2007-58-0015
Record Dates: First submitted 2018-02-15; First posted 2018-04-05 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Malnutrition
Keywords: Hospital readmissions; Seniors
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group
  Individual nutritional therapy
  Interventions: Dietary Supplement: Individual nutritional therapy
- Control (No Intervention): Control group
  Standard treatment

INTERVENTIONS:
Dietary Supplement: Individual nutritional therapy — Guidance from a clinical dietician.
  Individual nutrition plan
  A package containing foods and drinks, which will cover their nutritional needs the first day after discharge.
  A goodiebag containing samples on protein-rich milk-based drinks.
  Telephone follow-up after 4 and 30 days and the possibility to call the dietician in case of questions about nutrition.
  Arms: Intervention

SUMMARY:
The study is a randomized controlled study, ongoing over 16 weeks. At discharge, the intervention group receives guidance from a clinical dietician, where an individual nutrition plan is made. The dietitian will perform a telephone follow-up after 4 and 30 days. It will also be possible for the participant, relatives or municipality to contact the dietician if nutritional questions arise.

At the time of discharge the intervention group will receive a package containing foods and drinks that will cover their nutritional needs the first day after discharge.

They will also get a goodiebag containing samples on protein-rich milk-based drinks. Data is collected on quality of life, appetite, physical function, dietary intake, weight, height, energy and protein needs, as well as experience of discharge and cooperation with the municipality.

If there is a need, information about nutrition status will be sent to the municipality so the municipality can take over nutritional treatment.

The control group receives standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Oncology, Gastro-medical / Surgical, and Medical Department, HGH, Herlev.
* Age: 50+
* At admission, found in nutritional risk score ≥3 according to NRS-2002.
* On special food concept, Herlev's Glories during hospitalization
* Discharged to own home in a municipality in Planområde Midt (Ballerup, Herlev, Lyngby-Tårbæk, Gentofte, Gladsaxe, Rødovre, Egedal, Rudersdal, Furesø).
* Can read, hear and understand Danish
* Cognitive able to participate in the study, based on whether they are informed in time, place and own data.

Exclusion Criteria:

* Food allergy or intolerance
* Planned weight loss or following a special diet
* Receives enteral or parenteral nutrition
* Patients with moderate to severe dysphagia, defined with a need for gratin or a creamy diet
* Patients who does not want a food package or goodiebag
* Patients who are permanently bedridden
* Patients who are discharged to nursing homes or rehabilitation
* Patients in isolation
* Late palliative patients
* Terminal patients

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Hospital readmissions | 6 months

SECONDARY OUTCOMES:
Mortality | 30 days, 16 weeks, 6 months
Weight | 16 weeks
Protein intake | 16 weeks
  24 hour recall
Energi Intake | 16 weeks
  24 hour recall
Appetite | 16 weeks
  SNAQ
Health related Quality of life | 16 weeks
  EQ-5D
Physical function | 16 weeks
  30-s CST
Hospital readmissions | 30 days, 16 weeks
Combined adverse advents | 30 days, 16 weeks, 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Unit for Dietetics and Nutrition Research, Herlev hosipital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munk T, Svendsen JA, Knudsen AW, Ostergaard TB, Thomsen T, Olesen SS, Rasmussen HH, Beck AM. A multimodal nutritional intervention after discharge improves quality of life and physical function in older patients - a randomized controlled trial. Clin Nutr. 2021 Nov;40(11):5500-5510. doi: 10.1016/j.clnu.2021.09.029. Epub 2021 Sep 24. PMID 34656032
- [Derived] Munk T, Svendsen JA, Knudsen AW, Ostergaard TB, Beck AM. Effect of nutritional interventions on discharged older patients: study protocol for a randomized controlled trial. Trials. 2020 Apr 28;21(1):365. doi: 10.1186/s13063-020-04301-6. PMID 32345358